CLINICAL TRIAL: NCT01044693
Title: Effect of Nebivolol on Blood Pressure in a Model of Hypertension Sensitive to Potentiation of Nitric Oxide Bioactivity
Brief Title: Nebivolol in the Supine Hypertension of Autonomic Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 091252
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension; Pure Autonomic Failure; Multiple System Atrophy
Keywords: supine Hypertension; autonomic failure; nitric oxide; nebivolol
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure; Multiple System Atrophy | interventions — Sugars; Nebivolol; Metoprolol; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo capsule (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo
- Nebivolol 5 mg (Experimental): Nebivolol 5 mg capsule
  Interventions: Drug: Nebivolol 5 mg
- Metoprolol tartrate 50 mg (Active Comparator): Metoprolol tartrate 50 mg single oral dose
  Interventions: Drug: metoprolol tartrate 50 mg
- Sildenafil 25 mg (Active Comparator): Sildenafil 25 mg single oral dose
  Interventions: Drug: Sildenafil25 mg

INTERVENTIONS:
Drug: Placebo — Placebo capsule
  Other Names: sugar pill
  Arms: Placebo capsule
Drug: Nebivolol 5 mg — Nebivolol 5mg single oral dose
  Other Names: Bystolic
  Arms: Nebivolol 5 mg
Drug: metoprolol tartrate 50 mg — metoprolol tartrate 50 mg single oral dose
  Other Names: Lopressor
  Arms: Metoprolol tartrate 50 mg
Drug: Sildenafil25 mg — Sildenafil 25 mg single oral dose
  Other Names: Viagra
  Arms: Sildenafil 25 mg

SUMMARY:
The purpose of this study is to evaluate the effect of the antihypertensive drug, nebivolol (Bystolic), compared to metoprolol (Lopressor) and sildenafil (Viagra) on blood pressure in patients with autonomic failure and supine hypertension.

DETAILED DESCRIPTION:
Nebivolol is distinct among beta-blockers by its ability to increase nitric oxide (NO) bioactivity. The contribution of this effect to the pharmacological actions of the drug, however, is difficult to ascertain in normal subjects because of the confounding contribution of the autonomic nervous system. Autonomic failure patients provide a unique model of hypertension devoid of autonomic modulation but sensitive to NO mechanisms. We propose to determine the effect of nebivolol on blood pressure in this patient population. A decrease in blood pressure will imply increased bioactivity of NO. Comparisons will be made with placebo, metoprolol (as a negative control) and sildenafil (as a positive control).

ELIGIBILITY:
Inclusion Criteria:

* Male or female and aged 18 years or over.
* Clinical diagnosis of orthostatic hypotension associated with Primary Autonomic Failure (Parkinson Disease, Multiple System Atrophy and Pure Autonomic Failure).
* A documented fall in systolic blood pressure of at least 20 mmHg, or in diastolic blood pressure of at least 10 mmHg, within 3 minutes after standing.
* Supine hypertension, defined as a systolic blood pressure >150 mm Hg or diastolic blood pressure > 90 mm Hg.
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.

Exclusion Criteria:

* Have changed dose, frequency and or type of prescribed medication, within two weeks of study start.
* Women of childbearing potential who are not using a medically accepted contraception.
* Have, in the investigator's opinion, any significant cardiac, systemic, hepatic, or renal illness.
* Diabetes mellitus or insipidus.
* In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing.
* In the investigator's opinion, are unable to adequately co-operate because of individual or family situation.
* In the investigator's opinion, are suffering from a mental disorder that interferes with the diagnosis and/or with the conduct of the study, e.g. schizophrenia, major depression, dementia.
* Are not able or willing to comply with the study requirements for the duration of the study.
* Persons on drugs with beta-blocking potential (e.g., amiodarone), persons taking scheduled or as needed nitrates and persons on drugs with alpha-blocking potential (e.g. tamsulosin).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Biaggioni I, Garcia F, Inagami T, Haile V. Hyporeninemic normoaldosteronism in severe autonomic failure. J Clin Endocrinol Metab. 1993 Mar;76(3):580-6. doi: 10.1210/jcem.76.3.7680352.
- [Background] Cockcroft JR, Chowienczyk PJ, Brett SE, Chen CP, Dupont AG, Van Nueten L, Wooding SJ, Ritter JM. Nebivolol vasodilates human forearm vasculature: evidence for an L-arginine/NO-dependent mechanism. J Pharmacol Exp Ther. 1995 Sep;274(3):1067-71. PMID 7562470
- [Background] Gamboa A, Shibao C, Diedrich A, Paranjape SY, Farley G, Christman B, Raj SR, Robertson D, Biaggioni I. Excessive nitric oxide function and blood pressure regulation in patients with autonomic failure. Hypertension. 2008 Jun;51(6):1531-6. doi: 10.1161/HYPERTENSIONAHA.107.105171. Epub 2008 Apr 21. PMID 18426998
- [Background] Gupta S, Wright HM. Nebivolol: a highly selective beta1-adrenergic receptor blocker that causes vasodilation by increasing nitric oxide. Cardiovasc Ther. 2008 Fall;26(3):189-202. doi: 10.1111/j.1755-5922.2008.00054.x. PMID 18786089
- [Background] Shannon J, Jordan J, Costa F, Robertson RM, Biaggioni I. The hypertension of autonomic failure and its treatment. Hypertension. 1997 Nov;30(5):1062-7. doi: 10.1161/01.hyp.30.5.1062. PMID 9369256
- [Background] Tzemos N, Lim PO, MacDonald TM. Nebivolol reverses endothelial dysfunction in essential hypertension: a randomized, double-blind, crossover study. Circulation. 2001 Jul 31;104(5):511-4. doi: 10.1161/hc3001.094207. PMID 11479245

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Metoprolol Then Sildenafil Then Nebivolol; Placebo Then Nebivolol Then Metoprolol Then Sildenafil; Placebo Then Sildenafil Then Nebivolol Then Metoprolol; Placebo Then Sildenafil Then Metoprolol Then Nebivolol; Nebivolol Then Placebo Then Metoprolol Then Sildenafil; Metoprolol Then Sildenafil Then Placebo Then Nebivolol; Sildenafil Then Nebivolol Then Placebo Then Metoprolol; Metoprolol Then Placebo Then Nebivolol Then Sildenafil; Nebivolol Then Metoprolol Then Sildenafil Then Placebo; Metoprolol Then Nebivolol Then Placebo Then Sildenafil; Metoprolol Then Sildenafil Then Nebivolol Then Placebo; Sildenafil Then Nebivolol Then Metoprolol Then Placebo; Sildenafil Then Metoprolol Then Nebivolol Then Placebo; Nebivolol Then Sildenafil Then Metoprolol Then Placebo; Nebivolol Then Placebo Then Sildenafil Then Metoprolol; Placebo Then Nebivolol Then Sildenafil Then Metoprolol: Single oral dose of: metoprolol tartrate 50 mg, sildenafil 25 mg, nebivolol 5 mg
Period: Overall Study
Arm/Group | Placebo Then Metoprolol Then Sildenafil Then Nebivolol | Placebo Then Nebivolol Then Metoprolol Then Sildenafil | Placebo Then Sildenafil Then Nebivolol Then Metoprolol | Placebo Then Sildenafil Then Metoprolol Then Nebivolol | Nebivolol Then Placebo Then Metoprolol Then Sildenafil | Metoprolol Then Sildenafil Then Placebo Then Nebivolol | Sildenafil Then Nebivolol Then Placebo Then Metoprolol | Metoprolol Then Placebo Then Nebivolol Then Sildenafil | Nebivolol Then Metoprolol Then Sildenafil Then Placebo | Metoprolol Then Nebivolol Then Placebo Then Sildenafil | Metoprolol Then Sildenafil Then Nebivolol Then Placebo | Sildenafil Then Nebivolol Then Metoprolol Then Placebo | Sildenafil Then Metoprolol Then Nebivolol Then Placebo | Nebivolol Then Sildenafil Then Metoprolol Then Placebo | Nebivolol Then Placebo Then Sildenafil Then Metoprolol | Placebo Then Nebivolol Then Sildenafil Then Metoprolol
Started | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Completed | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with primary forms of autonomic failure and supine hypertension
Groups:
- All Study Participants: Participants who were randomized to receive placebo, metoprolol, sildenafil and nebivolol in any order
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.6 (3.2)
Duration of disease [Mean (Standard Deviation); unit: years] | 8 (6)
Diagnosis [Number; unit: participants]
  Pure autonomic failure | 10
  Parkinson Disease with autonomic failure | 4
  Multiple System Atrophy | 6
Medical history of essential hypertension [Number; unit: participants]
  yes | 4
  No | 16
Systolic BP, supine [Mean (Standard Deviation); unit: mm Hg] | 169 (24)
Systolic BP, upright [Mean (Standard Deviation); unit: mm Hg] | 83 (25)
Heart rate, supine [Mean (Standard Deviation); unit: bpm] | 68 (10)
Heart rate, upright [Mean (Standard Deviation); unit: bpm] | 83 (15)
Plasma norepinephrine, supine [Mean (Standard Deviation); unit: pg/mL] | 136 (98)
Plasma norepinephrine, upright [Mean (Standard Deviation); unit: pg/mL] | 253 (209)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure During the Night
Description: Maximal change from baseline in systolic blood pressure, measured from 8 pm to 8 am, after a single dose of the intervention
Time Frame: 8 pm - 8 am
Population: Participants who completed the 4 treatment arms
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo Capsule | Nebivolol 5 mg | Metoprolol Tartrate 50 mg | Sildenafil 25 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
mm Hg
  Baseline supine at 8 pm | 154 (7) | 162 (5) | 157 (5) | 158 (6)
  Change in systolic BP | 1 (7) | -24 (9) | -7 (6) | -20 (6)
Statistical Analysis 1: Comparison: Placebo Capsule vs Nebivolol 5 mg; The main comparisons were between the active treatment groups versus placebo. We hypothesized that if NO-mediated vasodilation contributes to the BP-lowering effect of nebivolol then BP will be lowered by nebivolol and sildenafil, but not by metoprolol in autonomic failure patients; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo Capsule vs Sildenafil 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo Capsule vs Metoprolol Tartrate 50 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis

2. Secondary Outcome: Nocturnal Urinary Sodium Excretion
Description: Nocturnal sodium excretion was defined as the ratio of urinary sodium to urinary creatinine.
Time Frame: 8 pm - 8 am
Population: Participants with complete urine collections during the 4 study nights
Measure: Mean (Standard Error); unit: mEq/mg
Arm/Group | Placebo Capsule | Nebivolol 5 mg | Metoprolol Tartrate 50 mg | Sildenafil 25 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14
mEq/mg | 0.145 (0.015) | 0.127 (0.011) | 0.139 (0.019) | 0.125 (0.018)
Statistical Analysis 1: Comparison: Placebo Capsule vs Nebivolol 5 mg vs Metoprolol Tartrate 50 mg vs Sildenafil 25 mg; The main comparisons were between the active treatment groups versus placebo; Test type: Superiority or Other; p = 0.607, ANOVA

3. Secondary Outcome: Orthostatic Tolerance the Following Morning
Description: Orthostatic tolerance was defined as the area under the curve of standing systolic blood pressure calculated by the trapezoidal rule (upright systolic blood pressure multiplied by standing time) during a 10-minute standing test
Time Frame: 10 min standing
Population: Comparisons were made only for patients who could stand after all treatment groups
Measure: Mean (Standard Error); unit: mm Hg*min
Arm/Group | Placebo Capsule | Nebivolol 5 mg | Metoprolol Tartrate 50 mg | Sildenafil 25 mg
Number analyzed (Participants) | 11 | 11 | 11 | 11
mm Hg*min | 594 (108) | 675 (113) | 696 (128) | 575 (106)
Statistical Analysis 1: Comparison: Placebo Capsule vs Nebivolol 5 mg vs Metoprolol Tartrate 50 mg vs Sildenafil 25 mg; The main comparisons were between the active treatment groups versus placebo; Test type: Superiority or Other; p = 0.597, ANOVA

4. Secondary Outcome: Change in Heart Rate During the Night
Description: Change from baseline (8 pm) in heart rate at the time of maximal BP-lowering effect
Time Frame: 8 pm - 8 am
Population: Participants who completed the 4 treatment arms
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Placebo Capsule | Nebivolol 5 mg | Metoprolol Tartrate 50 mg | Sildenafil 25 mg
Number analyzed (Participants) | 20 | 20 | 20 | 20
bpm | -3 (2) | -6 (2) | -6 (2) | 0 (2)
Statistical Analysis 1: Comparison: Nebivolol 5 mg vs Metoprolol Tartrate 50 mg; The main comparisons were between the negative chronotropic effect of nebivolol and metoprolol at the time when BP-lowering effects were maximal; Test type: Superiority or Other; p = 0.996, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 day for each intervention
Description: Safety population included all participants
Arm/Group | Placebo Capsule | Nebivolol 5 mg | Metoprolol Tartrate 50 mg | Sildenafil 25 mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Capsule (N=20) | Nebivolol 5 mg (N=20) | Metoprolol Tartrate 50 mg (N=20) | Sildenafil 25 mg (N=20)
fall (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant got up on his own to go to the bathroom during the night, partly falling and injuring his right 5th finger (dislocated).
Urinary Tract Infection and diarrhea (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — During study participation, it was found that she had a urinary tract infection (UTI), which contributed to the worsening of hypotension. Subject was taken off the study and treatment for UTI started. She was discharged without further incident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No